CLINICAL TRIAL: NCT06179524
Title: Phase II Clinical Study of CAR-T-19 Injection in the Treatment of CD19-positive Relapsed/refractory B-cell Acute Lymphoblastic Leukemia(B-ALL) Under 25 Years of Age (inclusive)
Brief Title: CAR-T-19 Injection in the Treatment of CD19-positive Relapsed/Refractory B-ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Yongtai Ruike Biotechnology Company Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT19-ALL-02
Record Dates: First submitted 2023-12-01; First posted 2023-12-22 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Relapsed B-cell Acute Lymphoblastic Leukemia; Refractory B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T-19 cells (Experimental): CAR-T-19 cells injection: 2.5 x10^6 cells/kg（range 0.8-2.5×10^6 cells/kg）
  Interventions: Biological: CAR-T-19 cell injection

INTERVENTIONS:
Biological: CAR-T-19 cell injection — The functional component of CAR-T-19 cell injection is T cells that have been genetically modified to express anti CD19 chimeric antigen receptors.

SUMMARY:
This is a phase II clinical study to evaluate the safety and efficacy of CAR-T-19 injection in the treatment of CD19-positive relapsed/refractory B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
This is a multiple-center, single-arm, open-label study. After meeting the eligibility criteria and enrolling on the trial, patients will undergo leukapheresis for collection of autologous lymphocytes, patients will then proceed to lymphodepleting chemotherapy with cyclophosphamide 300mg/m^2 and fludarabine 30mg/m^2 for 3 consecutive days followed by the infusion of CD19 CAR T-cells at a target dose of 2.5 x10^6 cells/kg（range 0.8-2.5×10^6 cells/kg）.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in clinical trial, The Participants or his legal guardian is fully understands this clinical trial and signs the Informed Consent Form (ICF); Willing to follow and be able to complete all trial procedures.
2. Age≤25 years old at the time of screening, regardless of gender.
3. Bone marrow examination confirmed the diagnosis of B-ALL, and meet one of the following conditions： Relapsed B-ALL：1）Relapse within 12 months of the first remission；2）Recurrence occurring again more than 12 months after the first remission,, relapsed or not responded after first-line/multi-line salvage chemotherapy；3) Experienced two or more bone marrow recurrences; 4） recurrence after autologous or allogeneic hematopoietic stem cell transplantation； Refractory B-ALL：1）failed to achieve complete remission after 2 cycles of standard induction chemotherapy.
4. Ph+ALL patients are eligible：1）Relapsed or refractory after receiving at least two Tyrosine kinase inhibitors (TKI) treatments；If Ph+ALL patients with t315i mutation are resistant to first- and second-generation TKIs, in the absence of effective TKI therapy, patients are not required to receive at least two TKIs；2）cannot tolerate TKI treatment；3）Presence of contraindications to TKI therapy.
5. Bone marrow (BM) or peripheral blood (PB) tumor cells were measured to express CD19 at screening.
6. Bone marrow blasts ≥ 5% at screening.
7. Adequate organ function and must meet the following criteria： Alanine aminotransferase (ALT) ≤ 5 ×Upper limit of normal value(ULN)；Total serum bilirubin ≤ 2.0 ×ULN(（for Gilbert syndrome, total bilirubin≤3.0×ULN)；in non-oxygen state, No > grade 1 dyspnea, Blood oxygen saturation > 95%；left ventricular ejection fraction(LVEF) ≥ 50%；Serum creatinine≤1.5 × ULN；
8. Karnofsky（age≥16 years）performance status≥70 or Lansky（age<16 years）performance status≥50.
9. Life expectancy ≥ 12 weeks.
10. Adequate venous access (for apheresis) and no other contraindications to apheresis.
11. Negative blood/urine pregnancy test in women of childbearing potential before screening and within 3 days prior to cell infusion, and any male and female patients of childbearing potential must agree to use an effective method of contraception throughout the study and for at least 2 years after CAR-T-19 infusion. In the judgment of the investigator, a patient of childbearing potential means that he/she is biologically capable of having children and having a normal sexual life.
12. For Participants who have previously undergone allogeneic hematopoietic stem cell transplantation, CAR-T-19 cell preparation is performed using their previous donor peripheral blood， and the donor needs to meet the following conditions：1）Have donated bone marrow/hematopoietic stem cells as a transplant donor for the patient；2）Age ≥8 years at screening；3）Voluntary participation in clinical studies; the donor (and legal guardian, if applicable) am fully aware of and informed about this trial and have signed an informed consent form (ICF); Willing to follow and be able to complete all trial procedures；4）Have adequate venous access (for apheresis or venous blood collection) and no other contraindications to apheresis; 5) The etiological test results do not correspond to any of the exclusion criteria outlined in item 12. 6) Women of childbearing age have negative blood and urine pregnancy tests.7) Systemic glucocorticoid therapy is prohibited within one week prior to apheresis, with the exception of physiologically replacement doses of glucocorticoids (0.5 mg/kg/day of prednisone or equivalent doses of other corticosteroids).8) There are no cases of uncontrolled fungal, bacterial, viral, or other infections requiring intravenous treatment.

Exclusion Criteria:

1. Isolated extra-medullary disease relapse .
2. Participants with genetic syndromes, Patients with Down Syndrome will not be excluded.
3. Participants with Burkitt's lymphoma/leukemia.
4. Participants with active central nervous system disease.
5. Active central nervous system leukemia at screening(Defined as CNS-3 and CNS-2 grades with neurological symptoms as defined by NCCN guidelines and judged by the investigator to be active central leukemia).
6. Participants with a history of other malignant tumors or other malignant tumors at the same time (excluding fully treated cervical carcinoma in situ, basal cell or squamous epithelial cell skin cancer, local prostate cancer after radical resection, thyroid cancer, ductal carcinoma in situ after radical resection).
7. have or suspected to have fungal, bacterial, viral or other infections that are uncontrollable or require intravenous treatment.
8. Participants who have received HSCT within 3 months before screening or Presence of grade 2 to 4 active graft-versus-host disease (GVHD), and those who have received systemic drug therapy for GVHD within 4 weeks before infusion.
9. Received the following anti-tumor therapy before apheresis：1）Received any chemotherapy, targeted therapy, etc. within 4 weeks or at least 5 half-lives (whichever is shorter)；2）Radiotherapy within 14 days；3）Intrathecal treatment within 7 days；4) Received a donor lymphocyte transfusion (DLI) within 4 weeks; 5)Received Blinatumomab within 14 days.
10. Participants who have been treated with systemic glucocorticoids within 1 week before apheresis, physiological replacement doses of steroids are allowed.
11. Long-acting G-CSF is prohibited within 21 days and short-acting G-CSF is prohibited within 7 days before apheresis.
12. Any of the following applies:1）Hepatitis B surface antigen (HBsAg) positive or HBV-DNA quantity is higher than the upper limit of normal value；2）Hepatitis C virus antibody (HCV Ab) is positive and HCV RNA quantification is higher than the upper limit of normal values;3）Positive for human immunodeficiency virus antibody (HIV-Ab);4）EB virus DNA quantification is higher than the upper limit of normal values;5）Cytomegalovirus DNA quantification is higher than the upper limit of normal values.
13. Those who have received CAR-T therapy with any target.
14. Allergy to albumin and aminoglycoside antibiotics.
15. Received live vaccine within 6 weeks before screening.
16. Participants after organ transplantation (except hematopoietic stem cell transplantation).
17. participated in other interventional clinical studies (received active trial drug treatment) within 3 months before screening, or intend to participate in another clinical trial or receive another anti-tumor therapy.
18. Other investigators deem it inappropriate to participate in the study.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | 3 months
  ORR included complete response (CR) and CR with incomplete blood count recovery (CRi) as determined by an Independent Review Committee（IRC） assessment.

SECONDARY OUTCOMES:
ORR | 3 months
  ORR at 3 months after CAR-T-19 infusion as assessed by investigator.
ORR | 28 days
  ORR at 28 days after CAR-T-19 infusion as assessed by IRC and investigator.
Minimal residual disease（MRD） | 3 months
  MRD-negative ORR as assessed by Independent Review Committee (IRC) and investigator.
Best overall response (BOR) | 2 years
  BOR as assessed by Independent Review Committee (IRC) and investigator.
Duration of response (DOR) | 2 years
  DOR as assessed by Independent Review Committee (IRC) and investigator.
Event Free Survival（EFS） | 2 years
  EFS as assessed by Independent Review Committee (IRC) and investigator.
Recurrence Free Survival（RFS） | 2 years
  RFS as assessed by Independent Review Committee (IRC) and investigator.
Overall survival (OS) | 2 yeas
  Overall survival means the time from infusion of CAR-T-19 cells to death of participants from any cause.
AE safety | 2 years
  Number of participants with Adverse event (AE).
SAE safety | 2 years
  Number of participants with Serious adverse event (SAE)
ADA safety | 2 years
  Number of participants with Anti-drug antibody(ADA).
RCL safety | 15 years
  Number of participants with Replication Competent Lentivirus (RCL).
Pharmacokinetics (PK) Parameter-Cmax | 2 years
  Cmax
Pharmacokinetics (PK) Parameter-Tmax | 2 years
  Tmax
Pharmacokinetics (PK) Parameter-AUC0-t | 2 years
  AUC0-t
Pharmacokinetics (PK) Parameter- AUC0-28d | 2 years
  AUC0-28d
Pharmacokinetics (PK) Parameter- t1/2 | 2 years
  t1/2
Pharmacodynamics | 2 years
  The degree of clearance of CD19-positive B cells at different blood collection time points after cell infusion.
Serum cytokines-Interleukin 6 | 28 days
  The concentration levels of Interleukin 6（ IL-6）at each time point .
Serum cytokines-Interleukin 10 | 28 days
  The concentration levels of Interleukin 10（ IL-10）at each time point .
Serum cytokines-TNF-α | 28 days
  The concentration levels of tumor necrosis factor -α（ TNF-α） at each time point .
Serum cytokines-INF-γ | 28 days
  The concentration levels of Interferon -γ（INF-γ） at each time point .

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Zhu, Principal Investigator — Hematology Hospital of the Chinese Academy of Medical Sciences
Locations (1):
- Hematology Hospital of the Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: No